CLINICAL TRIAL: NCT01844037
Title: Renal Denervation Using the OneShot Ablation System
Brief Title: OneShot Renal Denervation Registry
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP1002
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Hypertension; Heart Failure; Diabetes Mellitus; Sleep Apnea
MeSH Terms: conditions — Hypertension; Heart Failure; Diabetes Mellitus; Sleep Apnea Syndromes

ARMS (1):
- Renal denervation (Other): Patients will be treated with the OneShot ablation system
  Interventions: Device: OneShot Ablation System

INTERVENTIONS:
Device: OneShot Ablation System — Renal denervation

SUMMARY:
This is a multi-center, prospective registry designed to monitor the outcomes of renal denervation with the OneShot Device in a real-world patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patient is an acceptable candidate for renal denervation based upon the Instructions for Use.
* Patient is ≥ 18 years old.
* Patient provided written informed consent.

Exclusion Criteria:

* Patients who are pregnant, nursing, or planning to become pregnant.
* Patients who have only one functioning kidney.
* Allergy to contrast or known hypersensitivity to device materials
* Patients with renal arteries < 4 mm in diameter.
* Patients whose life expectancy is less than the planned period of study involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in office systolic blood pressure (SBP) from baseline to 6 months | 6 months

SECONDARY OUTCOMES:
Acute procedural safety, defined as freedom from renal artery dissection or perforation requiring intervention. | One Week
Change in office diastolic blood pressure (DBP) | 6 and 12 months post procedure
Change in office SBP | 6 and 12 months post procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital San Raffaele, Milan, Italy